CLINICAL TRIAL: NCT05170061
Title: Ambulatory 24-Hour Cardiac Oxygen Consumption and Blood Pressure-Heart Rate Variability: Effects of Nebivolol and Valsartan Alone and in Combination
Brief Title: 24 Hour Ambulatory Cardiac Oxygen Consumption
Acronym: ACRPP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, JOSEPH IZZO, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BYS-IT-76
Record Dates: First submitted 2014-12-22; First posted 2021-12-27 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Hypertension
Keywords: Myocardial oxygen consumption; Systolic blood pressure; Diastolic blood pressure; Variability in hemodynamic indicators; Valsartan; Nebivolol; IEM ambulatory monitoring
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Valsartan

STUDY DESIGN:
Intervention Model Description: Random-order-entry 3-way crossover of active treatments; all participants receive all 3 active treatments with 6 possible experimental sequences (arms)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded: drugs formulated into capsules by an outside research pharmacist who held the codes until study completion
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Sequence 1: Nebivolol first, then valsartan, then combination of nebivolol/valsartan (Active Comparator): Nebivolol, 20 mg daily for 1 week followed by 40 mg daily for 3 weeks, followed by 1 week down-titration to 20 mg daily; then Valsartan, 160 mg daily for 1 week followed by 320 mg daily for 3 weeks, followed by 1-week down-titration to 160 mg daily; then Combination of nebivolol/valsartan 20/160 mg daily for 1 week followed by 40/320 mg daily for 3 weeks, followed by 1-week down-titration to 20/160 mg daily
  Interventions: Drug: Nebivolol; Drug: Valsartan; Drug: Nebivolol/valsartan combination
- Sequence 2: Nebivolol first, then combination of nebivolol/valsartan; then valsartan (Active Comparator): Nebivolol, 20 mg daily for 1 week followed by 40 mg daily for 3 weeks, followed by 1 week down-titration to 20 mg daily; then combination of nebivolol/valsartan 20/160 mg daily for 1 week followed by 40/320 mg daily for 3 weeks, followed by 1-week down-titration to 20/160 mg daily; then Valsartan, 160 mg daily for 1 week followed by 320 mg daily for 3 weeks, followed by 1-week down-titration to 160 mg daily
  Interventions: Drug: Nebivolol; Drug: Valsartan; Drug: Nebivolol/valsartan combination
- Sequence 3: Valsartan first, then Nebivolol, then combination of nebivolol/valsartan, (Active Comparator): Valsartan, 160 mg daily for 1 week followed by 320 mg daily for 3 weeks, followed by 1-week down-titration to 160 mg daily; then Nebivolol, 20 mg daily for 1 week followed by 40 mg daily for 3 weeks, followed by 1 week down-titration to 20 mg daily; then combination of nebivolol/valsartan 20/160 mg daily for 1 week followed by 40/320 mg daily for 3 weeks, followed by 1-week down-titration to 20/160 mg daily;
  Interventions: Drug: Nebivolol; Drug: Valsartan; Drug: Nebivolol/valsartan combination
- Sequence 4: Valsartan first, then combination of nebivolol/valsartan, then Nebivolol, (Active Comparator): Valsartan, 160 mg daily for 1 week followed by 320 mg daily for 3 weeks, followed by 1-week down-titration to 160 mg daily; then combination of nebivolol/valsartan 20/160 mg daily for 1 week followed by 40/320 mg daily for 3 weeks, followed by 1-week down-titration to 20/160 mg daily; then Nebivolol, 20 mg daily for 1 week followed by 40 mg daily for 3 weeks, followed by 1 week down-titration to 20 mg daily;
  Interventions: Drug: Nebivolol; Drug: Valsartan; Drug: Nebivolol/valsartan combination
- Sequence 5: Combination of nebivolol/valsartan first, then Nebivolol, then Valsartan, (Active Comparator): Combination of nebivolol/valsartan 20/160 mg daily for 1 week followed by 40/320 mg daily for 3 weeks, followed by 1-week down-titration to 20/160 mg daily; then Nebivolol, 20 mg daily for 1 week followed by 40 mg daily for 3 weeks, followed by 1 week down-titration to 20 mg daily; then Valsartan, 160 mg daily for 1 week followed by 320 mg daily for 3 weeks, followed by 1-week down-titration to 160 mg daily;
  Interventions: Drug: Nebivolol; Drug: Valsartan; Drug: Nebivolol/valsartan combination
- Sequence 6: Combination of nebivolol/valsartan first, then Valsartan, then Nebivolol, , (Active Comparator): Combination of nebivolol/valsartan 20/160 mg daily for 1 week followed by 40/320 mg daily for 3 weeks, followed by 1-week down-titration to 20/160 mg daily; then Valsartan, 160 mg daily for 1 week followed by 320 mg daily for 3 weeks, followed by 1-week down-titration to 160 mg daily; then Nebivolol, 20 mg daily for 1 week followed by 40 mg daily for 3 weeks, followed by 1 week down-titration to 20 mg daily; then
  Interventions: Drug: Nebivolol; Drug: Valsartan; Drug: Nebivolol/valsartan combination

INTERVENTIONS:
Drug: Nebivolol — Nebivolol 20 mg daily (1 week) followed by nebivolol 40 mg daily (3 weeks) followed by nebivolol 20 mg daily (1 week)
  Other Names: Bystolic
Drug: Valsartan — Valsartan 160 mg daily (1 week) followed by valsartan 320 mg daily (3 weeks) followed by valsartan 160 mg daily (1 week).
  Other Names: Diovan
Drug: Nebivolol/valsartan combination — Valsartan/Nebivolol, 160/20 mg daily (1 week) followed by valsartan/nebivolol 320/40 mg daily (3 weeks) followed by valsartan/nebivolol 160/20 mg daily (1 week)
  Other Names: Diovan/Bystolic

SUMMARY:
A randomized,double-blind, active controlled,15 week study to evaluate the effects of nebivolol and valsartan alone and in combination on 24-hour ambulatory cardiac work and variability of heart rate-mean central systolic pressure product.

DETAILED DESCRIPTION:
Subjects with hypertension (systolic blood pressure (SBP) >140 or diastolic blood pressure (DBP)>90, n=26) were studied using a double-blinded, forced-titration, sequence-controlled, crossover design with 3 experimental periods: Valsartan 320, nebivolol 40, and nebivolol/valsartan 320/40 mg daily. After 4 weeks of each drug, ambulatory pulse wave analysis (IEM MobilOGraph) was performed every 20 min for 24-hours. The primary hypothesis was that nebivolol/valsartan combination therapy would be superior to valsartan monotherapy in reducing mean 24-hour mean myocardial oxygen consumption determined by 24-hour ambulatory heart rate-central systolic pressure product [ACRPP]. A secondary hypothesis was that the combination would also reduce the variability of 24-hour myocardial oxygen consumption.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic hypertension, treated or untreated

  * Males and females, 18 years or older
  * Seated clinic systolic BP 145-184 mmHg inclusive or
  * Seated clinic diastolic BP 92-119 mmHg, inclusive.

Exclusion Criteria:

* Subjects with any of the following conditions will be excluded:

  * Any acute or chronic medical condition that, in the judgment of the investigator, renders the subject unable to complete the study, would interfere with optimal participation in the study, or cause significant risk to the subject
  * Concomitant or probable need for treatment with other cardiovascular or antihypertensive drugs that may affect blood pressure or influence the effects of study drugs, (e.g. NSAIDs, beta-agonist inhalers therapy for bronchospastic asthma, diuretics); other stable chronic medications that have little effect on study drugs (e.g. diabetes medications, hormone replacements, chronic pain medications. osteoporosis drugs, vitamins, cholesterol drugs, etc.) are permitted if continued at stable doses throughout study.
  * History of clinically significant adverse events with beta-blocker or angiotensin-receptor blocker
  * Known or suspected secondary hypertension (e.g., renovascular hypertension, primary hyperaldosteronism, etc.)
  * Known ischemic heart disease requiring continuous beta-blocker therapy (includes angina, prior transmural myocardial infarction, coronary artery bypass graft surgery or percutaneous transluminal coronary angioplasty or stenting within 6 months prior to study entry).
  * Dilated cardiomyopathy (NYHA Functional Class III-IV)
  * Clinically significant valvular heart disease or obstructive hypertrophic cardiomyopathy
  * Presence of clinically significant ventricular or supraventricular arrhythmias (e.g. atrial fibrillation/flutter), pre-excitation syndrome, second or third degree atrioventricular block, other conduction defects necessitating the implantation of a permanent cardiac pacemaker, or sick sinus syndrome.
  * Chronic kidney disease (serum creatinine >2.5 mg/dL)
  * Uncontrolled diabetes mellitus (hemoglobin A1c > 10%)
  * History of alcohol or other drug abuse within 6 months prior to enrollment
  * Positive pregnancy test or failure to practice adequate contraception in women of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Izzo, MD, Principal Investigator — SUNY Buffalo
Locations (1):
- Erie County Medical Center, Buffalo, New York, United States

REFERENCES:
- [Result] Izzo JL Jr, Khan SU, Saleem O, Osmond PJ. Ambulatory 24-hour cardiac oxygen consumption and blood pressure-heart rate variability: effects of nebivolol and valsartan alone and in combination. J Am Soc Hypertens. 2015 Jul;9(7):526-35. doi: 10.1016/j.jash.2015.03.009. Epub 2015 Mar 28. PMID 26116459

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the practice of the investigator and by advertisement
Pre-assignment Details: Males and females, 18 years or older with chronic hypertension, treated or untreated, were eligible if their seated mean clinic systolic BP was 145-179 mm Hg, inclusive, or clinic diastolic BP 92-119 mm Hg, inclusive. Prior antihypertensive drug therapy was discontinued prior to randomization.
Groups:
- Sequence 1: Nebivolol, Valsartan, Combination Nebivolol/Valsartan: Nebivolol (20 mg daily for 1 week, then 40 mg daily for 3 weeks, then 20 mg daily for 1 week); Valsartan (160 mg daily for 1 week, then 320 mg daily for 3 weeks, then 160 mg daily for 1 week), then Combination nebivolol/valsartan (20/160 mg daily for 1 week, then 40/320 mg daily for 3 weeks, then 20/160 mg daily for 1 week).
- Sequence 2: Nebivolol, Combination Nebivolol/Valsartan, Valsartan: Nebivolol (20 mg daily for 1 week, then 40 mg daily for 3 weeks, then 20 mg daily for 1 week); Combination nebivolol/valsartan (20/160 mg daily for 1 week, then 40/320 mg daily for 3 weeks, then 20/160 mg daily for 1 week); Valsartan (160 mg daily for 1 week, then 320 mg daily for 3 weeks, then 160 mg daily for 1 week)
- Sequence 3: Valsartan, Nebivolol, Combination Nebivolol/Valsartan: Valsartan (160 mg daily for 1 week, then 320 mg daily for 3 weeks, then 160 mg daily for 1 week); Nebivolol (20 mg daily for 1 week, then 40 mg daily for 3 weeks, then 20 mg daily for 1 week), Combination nebivolol/valsartan (20/160 mg daily for 1 week, then 40/320 mg daily for 3 weeks, then 20/160 mg daily for 1 week).
- Sequence 4: Valsartan, Combination Nebivolol/Valsartan, Nebivolol: Valsartan (160 mg daily for 1 week, then 320 mg daily for 3 weeks, then 160 mg daily for 1 week); Combination nebivolol/valsartan (20/160 mg daily for 1 week, then 40/320 mg daily for 3 weeks, then 20/160 mg daily for 1 week); Nebivolol (20 mg daily for 1 week, then 40 mg daily for 3 weeks, then 20 mg daily for 1 week),
- Sequence 5: Combination Nebivolol/Valsartan, Nebivolol, Valsartan: Combination nebivolol/valsartan (20/160 mg daily for 1 week, then 40/320 mg daily for 3 weeks, then 20/160 mg daily for 1 week); Nebivolol (20 mg daily for 1 week, then 40 mg daily for 3 weeks, then 20 mg daily for 1 week); Valsartan (160 mg daily for 1 week, then 320 mg daily for 3 weeks, then 160 mg daily for 1 week);
- Sequence 6: Combination Nebivolol/Valsartan, Valsartan, Nebivolol: Combination nebivolol/valsartan (20/160 mg daily for 1 week, then 40/320 mg daily for 3 weeks, then 20/160 mg daily for 1 week); Valsartan (160 mg daily for 1 week, then 320 mg daily for 3 weeks, then 160 mg daily for 1 week); Nebivolol (20 mg daily for 1 week, then 40 mg daily for 3 weeks, then 20 mg daily for 1 week),
Period: Overall Study
Arm/Group | Sequence 1: Nebivolol, Valsartan, Combination Nebivolol/Valsartan | Sequence 2: Nebivolol, Combination Nebivolol/Valsartan, Valsartan | Sequence 3: Valsartan, Nebivolol, Combination Nebivolol/Valsartan | Sequence 4: Valsartan, Combination Nebivolol/Valsartan, Nebivolol | Sequence 5: Combination Nebivolol/Valsartan, Nebivolol, Valsartan | Sequence 6: Combination Nebivolol/Valsartan, Valsartan, Nebivolol
Started | 5 | 5 | 4 | 4 | 4 | 4
Completed | 5 | 5 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence 1: Nebivolol, Valsartan, Nebivolol/Valsartan: Nebivolol, 20 mg daily for 1 week followed by 40 mg daily for 3 weeks, followed by 1 week down-titration to 20 mg daily; then Valsartan, 160 mg daily for 1 week followed by 320 mg daily for 3 weeks, followed by 1-week down-titration to 160 mg daily; then Combination of nebivolol/valsartan 20/160 mg daily for 1 week followed by 40/320 mg daily for 3 weeks, followed by 1-week down-titration to 20/160 mg daily
- Sequence 2: Nebivolol, Nebivolol/Valsartan, Valsartan: Nebivolol, 20 mg daily for 1 week followed by 40 mg daily for 3 weeks, followed by 1 week down-titration to 20 mg daily; then Combination of nebivolol/valsartan 20/160 mg daily for 1 week followed by 40/320 mg daily for 3 weeks, followed by 1-week down-titration to 20/160 mg daily; then Valsartan, 160 mg daily for 1 week followed by 320 mg daily for 3 weeks, followed by 1-week down-titration to 160 mg daily
- Sequence 3: Valsartan, Nebivolol, Nebivolol/Valsartan: Valsartan, 160 mg daily for 1 week followed by 320 mg daily for 3 weeks, followed by 1-week down-titration to 160 mg daily; then Nebivolol, 20 mg daily for 1 week followed by 40 mg daily for 3 weeks, followed by 1 week down-titration to 20 mg daily; then Combination of nebivolol/valsartan 20/160 mg daily for 1 week followed by 40/320 mg daily for 3 weeks, followed by 1-week down-titration to 20/160 mg daily
- Sequence 4: Valsartan, Nebivolol/Valsartan, Nebivolol: Valsartan, 160 mg daily for 1 week followed by 320 mg daily for 3 weeks, followed by 1-week down-titration to 160 mg daily; then Combination of nebivolol/valsartan 20/160 mg daily for 1 week followed by 40/320 mg daily for 3 weeks, followed by 1-week down-titration to 20/160 mg daily; then Nebivolol, 20 mg daily for 1 week followed by 40 mg daily for 3 weeks, followed by 1 week down-titration to 20 mg daily
- Sequence 5: Nebivolol/Valsartan, Nebivolol, Valsartan: Combination of nebivolol/valsartan 20/160 mg daily for 1 week followed by 40/320 mg daily for 3 weeks, followed by 1-week down-titration to 20/160 mg daily; then Nebivolol, 20 mg daily for 1 week followed by 40 mg daily for 3 weeks, followed by 1 week down-titration to 20 mg daily; then Valsartan, 160 mg daily for 1 week followed by 320 mg daily for 3 weeks, followed by 1-week down-titration to 160 mg daily
- Sequence 6: Nebivolol/Valsartan, Valsartan, Nebivolol: Combination of nebivolol/valsartan 20/160 mg daily for 1 week followed by 40/320 mg daily for 3 weeks, followed by 1-week down-titration to 20/160 mg daily; then Valsartan, 160 mg daily for 1 week followed by 320 mg daily for 3 weeks, followed by 1-week down-titration to 160 mg daily; then Nebivolol, 20 mg daily for 1 week followed by 40 mg daily for 3 weeks, followed by 1 week down-titration to 20 mg daily
- Total: Total of all reporting groups
Arm/Group | Sequence 1: Nebivolol, Valsartan, Nebivolol/Valsartan | Sequence 2: Nebivolol, Nebivolol/Valsartan, Valsartan | Sequence 3: Valsartan, Nebivolol, Nebivolol/Valsartan | Sequence 4: Valsartan, Nebivolol/Valsartan, Nebivolol | Sequence 5: Nebivolol/Valsartan, Nebivolol, Valsartan | Sequence 6: Nebivolol/Valsartan, Valsartan, Nebivolol | Total
Number analyzed (Participants) | 5 | 5 | 4 | 4 | 4 | 4 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 3 | 3 | 3 | 21
  >=65 years | 1 | 1 | 0 | 1 | 1 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10) | 56 (9) | 59 (10) | 57 (9) | 56 (11) | 59 (11) | 58 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 3 | 2 | 2 | 17
  Male | 1 | 2 | 1 | 1 | 2 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 3 | 4 | 4 | 4 | 23
  White | 1 | 1 | 1 | 0 | 0 | 0 | 3
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 4 | 4 | 4 | 4 | 26

OUTCOME MEASURES:

1. Primary Outcome: ACRPP: 24-hour Ambulatory Central Rate-pressure Product (Also Called TTI, CTTI)
Description: ACRPP is the product of estimated aortic mean systolic pressure (mean aortic pressure estimated using a transfer function applied to brachial cuff blood pressure) during the systolic time interval adjusted for heart rate. Units are (mmHg*beats/min).
Time Frame: measurement after 4 weeks in each treatment arm
Population: Each group represents total number who received that treatment arm (n=26) given randomly in 6 possible sequences: N-V-N/V, N-N/V-V, V-N-N/V, V-N/V-N, N/V-N-V, N/V-V-N) Design was used to minimize any potential carryover bias from prior treatment, in part because of the relatively short duration of each treatment and the absence of washout periods between arms.
Measure: Mean (Standard Deviation); unit: mmHg*beats/min
Groups:
- Nebivolol: Nebivolol, 20 mg daily for 1 week followed by 40 mg daily for 3 weeks, followed by 1 week down-titration to 20 mg daily
- Valsartan: Valsartan, 160 mg daily for 1 week followed by 320 mg daily for 3 weeks, followed by 1-week down-titration to 160 mg daily
- Nebivolol/Valsartan: Combination of nebivolol/valsartan 20/160 mg daily for 1 week followed by 40/320 mg daily for 3 weeks, followed by 1-week down-titration to 20/160 mg daily
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg*beats/min | 2531 (400) | 2824 (530) | 2484 (368)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; Sequential analysis: if the first analysis (paired t-test to determine superiority of nebivolol/valsartan over valsartan ) reached p< 0.05, the superiority of nebivolol over valsartan was tested (paired-t test); if the second comparison reached p < 0.05, the superiority of nebivolol/valsartan over nebivolol was tested (paired-t test); Test type: Superiority; p = 0.05, t-test, 2 sided — see above; paired analysis

2. Secondary Outcome: Cuff SBP
Description: Seated office cuff systolic blood pressure (mmHg)
Time Frame: After 4 weeks in each treatment arm
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg | 150 (17) | 148 (17) | 146 (20)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

3. Secondary Outcome: Cuff DBP
Description: Seated office cuff diastolic blood pressure (mmHg)
Time Frame: After 4 weeks in each treatment arm
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg | 84 (12) | 87 (13) | 81 (12)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

4. Secondary Outcome: Ambulatory Brachial Double Product
Description: 24-hour mean heart rate x 24-hour mean systolic BP
Time Frame: After 4 weeks in each treatment arm
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg*beats/min
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg*beats/min | 9329 (1572) | 11239 (2336) | 9154 (1607)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

5. Secondary Outcome: Ambulatory Mean Heart Rate
Description: Mean heart rate over 24 hours
Time Frame: After 4 weeks in each treatment arm
Population: all participants
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
beats/min | 64 (8) | 77 (16) | 63 (10)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

6. Secondary Outcome: Ambulatory Mean Central Diastolic BP
Description: Mean ambulatory aortic (central) diastolic pressure over 24 hours
Time Frame: After 4 weeks in each treatment arm
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg | 91 (13) | 90 (12) | 89 (13)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

7. Secondary Outcome: 24-hour Brachial Systolic BP
Description: Mean 24-hour ambulatory systolic BP
Time Frame: 4 weeks
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg | 147 (15) | 143 (16) | 145 (16)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

8. Secondary Outcome: 24-hour Brachial Diastolic BP
Description: Mean 24-hour ambulatory cuff diastolic BP
Time Frame: After 4 weeks in each treatment arm
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg | 89 (12) | 88 (12) | 87 (13)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

9. Secondary Outcome: Daytime ACRPP (Ambulatory Central Rate-Pressure Product (Also Called TTI, CTTI)
Description: Determined by ambulatory heart rate-central systolic pressure product during self-reported waking hours at the end of each study phase
Time Frame: After 4 weeks in each treatment arm
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg*beats/min
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg*beats/min | 2482 (368) | 2817 (394) | 2423 (390)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

10. Secondary Outcome: Nighttime ACRPP
Description: Determined by ambulatory heart rate-central systolic pressure product during self-reported sleeping hours
Time Frame: After 4 weeks in each treatment arm
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg*beats/min
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg*beats/min | 2454 (471) | 2564 (516) | 2309 (446)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

11. Secondary Outcome: Daytime Heart Rate
Description: Mean ambulatory heart rate during self-reported waking hours
Time Frame: After 4 weeks in each treatment arm
Population: all participants
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
beats/min | 64 (10) | 81 (13) | 64 (9)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

12. Secondary Outcome: Nighttime Heart Rate
Description: Mean ambulatory heart rate during self-reported sleeping hours
Time Frame: 4 weeks
Population: all participants
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
beats/min | 64 (9) | 74 (12) | 63 (10)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

13. Secondary Outcome: Daytime Central Systolic Pressure
Description: Mean ambulatory central systolic pressure during self-reported waking hours
Time Frame: After 4 weeks in each treatment arm
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg | 138 (11) | 135 (14) | 136 (14)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

14. Secondary Outcome: Nighttime Central Systolic Pressure
Description: Mean ambulatory central systolic pressure during self-reported sleeping hours
Time Frame: 4 weeks
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg | 135 (20) | 130 (19) | 131 (16)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

15. Secondary Outcome: Daytime Brachial Systolic Pressure
Description: Mean ambulatory brachial systolic pressure during self-reported waking hours
Time Frame: After 4 weeks in each treatment arm
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg | 149 (12) | 146 (15) | 147 (16)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

16. Secondary Outcome: Nighttime Brachial Systolic Pressure
Description: Mean ambulatory brachial systolic pressure during self-reported sleeping hours
Time Frame: 4 weeks
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg | 145 (21) | 138 (19) | 141 (17)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

17. Secondary Outcome: Daytime Central Diastolic Pressure
Description: Mean ambulatory central diastolic pressure during self-reported waking hours
Time Frame: 4 weeks
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg | 93 (11) | 93 (12) | 92 (13)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

18. Secondary Outcome: Nighttime Central Diastolic Pressure
Description: Mean ambulatory central diastolic pressure during self-reported sleeping hours
Time Frame: After 4 weeks in each treatment arm
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg | 89 (15) | 86 (15) | 85 (14)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority; p = 0.05, t-test, 2 sided

19. Secondary Outcome: Daytime Brachial Diastolic Pressure
Description: Mean ambulatory brachial diastolic pressure during self-reported waking hours
Time Frame: 4 weeks
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg | 91 (10) | 91 (11) | 89 (13)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

20. Secondary Outcome: Nighttime Brachial Diastolic Pressure
Description: Mean ambulatory brachial diastolic pressure during self-reported sleeping hours
Time Frame: After 4 weeks in each treatment arm
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg | 87 (16) | 83 (14) | 83 (14)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

21. Secondary Outcome: Ambulatory Daytime Brachial Rate-pressure Product
Description: Mean ambulatory heart rate x brachial systolic blood pressure product during self-reported waking hours
Time Frame: After 4 weeks in each treatment arm
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg*beats/min
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg*beats/min | 9528 (1530) | 11869 (2265) | 9335 (1607)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

22. Secondary Outcome: Ambulatory Nighttime Brachial Rate-pressure Product
Description: Mean ambulatory heart rate x brachial systolic blood pressure product during self-reported sleeping hours
Time Frame: After 4 weeks in each treatment arm
Population: all participants
Measure: Mean (Standard Deviation); unit: mmHg*beats/min
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
Number analyzed (Participants) | 26 | 26 | 26
mmHg*beats/min | 9284 (1920) | 10338 (2449) | 8830 (1827)
Statistical Analysis 1: Comparison: Nebivolol vs Valsartan vs Nebivolol/Valsartan; see primary dependent variable; Test type: Superiority — see primary dependent variable; p = 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 15 weeks for each participant; approximately 1-year for the study overall
Description: same definitions
Arm/Group | Nebivolol | Valsartan | Nebivolol/Valsartan
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26

LIMITATIONS AND CAVEATS:
Relatively small sample size limits extrapolation. Small number of non-blacks precludes racial stratification.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No